CLINICAL TRIAL: NCT01260792
Title: Validation and Norms for Attention Deficit/Hyperactivity Disorder Scales in Children and Adults. Description of Associated Factors.
Brief Title: Children and Parents With ADHD and Related Disorders
Acronym: ChiP-ARD
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 09-APN-02
Record Dates: First submitted 2010-12-14; First posted 2010-12-15 (Estimated); Last update posted 2012-03-26 (Estimated); Status verified 2009-09

CONDITIONS: General Population; TDAH; Children Aged 5 to 18 Years
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Children: Children between 5 and 18 years old.
  Interventions: Other: questionnaire
- Adults: Parents of children between 5 and 18 years old
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: questionnaire — The teachers or the professors complete questionnaires on the child on their behavior in classes
  Groups: Children
Other: Questionnaire — The parents complete a questionnaire on the behavior of their child and on their own behavior
  Groups: Adults

SUMMARY:
Almost all rating scales for Attention-Deficit/Hyperactivity Disorder (ADHD) are not validated in France. This clearly hampers the development of the diagnosis and the monitoring of patients but also research in this domain. This study is conceived to collect data in the general population of children aged from 4 to 18 years in public schools in the city of Nice.

Children are pseudo-randomly selected from classes of randomly selected schools in the city of Nice (France). Teachers fill out questionnaires using a dedicated secured website, and ask parents to fill out a similar set of questionnaires regarding their child's behaviour at home. Since ADHD has a strong genetic components, parents are also asked to fill out questionnaires regarding their own behaviour at adulthood and in childhood retrospectively.

Additionally, known factors related to ADHD and other disorders as well as other putative factors are tested in the epidemiologic study.

ELIGIBILITY:
Inclusion Criteria:

* Child known for the teacher for at least three months so that his evaluation Reflect most faithfully possible the usual behavior of the child,
* Child having the Frenchman for mother tongue to avoid the consequences on him Behavior of a linguistic obstacle,
* Authorization to use the data signed by at least one of the parents of the child and by the very child when he is old at least of six years.
* Parents speaking and reading the Frenchman.

Exclusion Criteria:

* Child known to follow a specific treatment of a disorder(confusion)attentional with / without Hyperactivity-impulsiveness (eg. Ritaline Ò, Ritaline Ò LP, Arranged Ò LP, Strattera Ò) Whatever is its duration. Indeed, a selection on this criterion would introduce a way Major which(who) would return the less reliable results(profits) of the study.
* Child presenting a known neurological or psychiatric disorder, or a deficit Intellectual because the attentional disorders(confusions), the psychomotor excitement and The impulsiveness can be symptoms inherent to the other pathologies Neurological and\or psychiatric.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Two non-independant study groups: children aged 5 to 18, and at least one of their parents
Sampling Method: Probability Sample
Enrollment: 2600 (Actual)
Dates: Start 2010-02; Primary Completion 2011-07 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Validity of studied instruments | at time=0
  The only criterion of evaluation towards the type of the study and its main objective is Validity of the studied instruments

CONTACTS AND LOCATIONS:
Overall Officials: Hervé CACI, PH, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (1):
- CHU de Nice, Nice, France

REFERENCES:
- [Derived] Caci HM, Morin AJ, Tran A. Prevalence and correlates of attention deficit hyperactivity disorder in adults from a French community sample. J Nerv Ment Dis. 2014 Apr;202(4):324-32. doi: 10.1097/NMD.0000000000000126. PMID 24647218
- [Derived] Morin AJ, Tran A, Caci H. Factorial Validity of the ADHD Adult Symptom Rating Scale in a French Community Sample: Results From the ChiP-ARD Study. J Atten Disord. 2016 Jun;20(6):530-41. doi: 10.1177/1087054713488825. Epub 2013 May 31. PMID 23729493
- [Derived] Caci HM, Morin AJ, Tran A. Teacher Ratings of the ADHD-RS IV in a Community Sample: Results From the ChiP-ARD Study. J Atten Disord. 2016 May;20(5):434-44. doi: 10.1177/1087054712473834. Epub 2013 Feb 19. PMID 23422236